CLINICAL TRIAL: NCT00211627
Title: Clinical Study to Determine Safety and Effectiveness of KEEPASLEEP Device in Simple Snorers.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miller, Chipp St. Kevin, M.D. (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MILC - KEEPASLEEP - 0704
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Snoring; Sleep Apnea Syndromes
MeSH Terms: conditions — Snoring; Sleep Apnea Syndromes

INTERVENTIONS:
Device: KEEPASLEEP enhanced breathing device

SUMMARY:
Study to demonstrate the safety and effectiveness of a new oral enhanced airway device to treat simple snoring.

DETAILED DESCRIPTION:
The Keepasleep airway device is a novel and unique buccopharyngeal airway device to enhance breathing during sleep. This method has not been described in the medical literature and has been successful in limited testing. This clinical trial is to determine the safety and effectiveness of the KEEPASLEEP device utilizing 30 subjects with simple snoring. Each subject will serve as his/her own control. The device augments airflow into the posterior pharynx to minimize airway collapse,tissue vibration, and consequent snoring.The device passes through the retromaxillary space and requires that the subject be absent their wisdom teeth.

ELIGIBILITY:
Inclusion Criteria:- 18 yrs. of age or greater

* generally good health
* Intact dentition / ABSENT upper and lower wisdom teeth ( by extraction or lack of development )
* Simple snoring( documented by observer) or mild sleep apnea RDI < 15 ( documented by polysomnogram)
* Subject must have a concerned observer to assess of sleep and snoring behavior during trial period

Exclusion Criteria:- Presence of Wisdom teeth (third molars)

* active oral disease
* acute illness
* BMI (body mass index) > 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Reduction/Elimination of snoring behavior

CONTACTS AND LOCATIONS:
Overall Officials: Chipp K. Miller, M.D., Principal Investigator — St. Johns Health Center
Locations (1):
- Chipp St. Kevin Miller M.D., Santa Monica, California, United States